CLINICAL TRIAL: NCT00428467
Title: Pronounced Apical Dilatation in Failing Left Ventricles - a New Option for Surgical Remodelling Techniques
Brief Title: Apical Compression Stitch - a New Option for LV Remodelling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Apex-stitch; 236/04
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Heart Failure; Left Ventrikular Remodelling; Left Ventricular Geometry
Keywords: Heart Failure; LV Geometry; Heart MRT
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Procedure: LV Apex Compression

SUMMARY:
The current study analyses the LV geometry of failing LVs measured by MRI scanning with respect to systolic versus diastolic function. A new surgical method for remodelling enlarged left ventricles is introduced.An apical remodelling stitch led to significant remodelling which was accompanied by improvement in ventricular function.

DETAILED DESCRIPTION:
Heart failure is a common disease and remains a growing cause of morbidity and mortality worldwide. The poor prognosis of dietetic and medical treatment has led to Increasing interest in interventional and surgical techniques for improvement of LV function.

Besides heart transplantation surgical interventions in heart failure patients focussed on mitral valve repair, biventricular stimulation and correction of coronary artery disease. A partial ventriculectomy as a true remodelling procedure has been invented by Battista with varying clinical results and reported high mortalities up to 20%. More commonly used is the Dor procedure , which is applicable for anterior wall aneurysms and has excellent short and long term results. On the other hand it has been designed for chronic aneurysms and is not suitable for dilated cardiomyopathies or subacute infarctions. More recently medical devices like the Acorn™ net or the Myosplint™ have been invented. Both require implantation of significant foreign material and are combined with inherent disadvantages. The Acorn™ device prevents progressive dilatation, but does not support systolic ventricular function, whereas the Myospilnt™ creates a less spherical geometry but not a physiological shape of the left ventricle (LV).

Detailed knowledge of the underlying geometrical changes in failing left ventricles is a prerequisite to achieve improvement in function by surgery . It has been described that with progressive heart failure, the oval form changes towards a more spherical geometry. To classify the shape and amount of deformation, several indices have been defined . The classical sphericity index (SI) as the ratio between the short and long axis is commonly used and is able to predict volume increases e.g. after myocardial infarctions . Furthermore, it has been used for evaluation of remodelling surgery and mitral valve repair in heart failure patients . This index serves well for an overall judgement of the left ventricular geometry, but does not pay attention to asymmetrical aspects of remodelling in heart failure, which is present e.g. after myocardial infarctions. Especially the apex is not considered sufficiently, although it can be reshaped ideally in procedures like the Dor operation . Therefore a focus on this region of the left ventricle is desirable from a surgical point of view.

Cine MRI scanning of the heart has gained increasing acceptance in the diagnosis of ventricular geometry changes , as it is highly accurate in determining global myocardial function without using ionising radiation or assumptions of ventricular shape , which are major drawbacks of other imaging modalities such as nuclear ventriculography or echocardiography , respectively.

The current study analyses the LV geometry of failing LVs measured by MRI scanning with respect to systolic versus diastolic function. A new surgical method for remodelling enlarged left ventricles is introduced.

ELIGIBILITY:
Inclusion Criteria:

* Gender
* Coronary Disease
* impaired LF Function (EF<35%)

Exclusion Criteria:

* Pacemaker
* emergency Case,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Omer Dzemali, MD, Principal Investigator — Dept. of Thoracic and Cardiovascular Surgery, J.W. Goethe University, Frankfurt am Main, Germany